CLINICAL TRIAL: NCT02461927
Title: Ketamine for The Rapid Treatment of Major Depression and Alcohol Use Disorder
Brief Title: Ketamine for the Rapid Treatment of Major Depressive Disorder and Alcohol Use Disorder
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MHBB-009-16F; GY 0002 (Other: VA Connecticut Healthcare System)
Record Dates: First submitted 2015-06-01; First posted 2015-06-03 (Estimated); Results first posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Major Depressive Disorder; Alcohol Use Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Alcoholism | interventions — Ketamine; Naltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Ketamine + Naltrexone (Experimental): Subjects in this arm will receive (1) intravenous ketamine treatment once a week for 4 weeks (a total of 4 infusions) with a follow-up of 4 weeks and (2) intramuscular naltrexone once a month (a total of 2 injections).
  Interventions: Drug: Ketamine + Naltrexone
- Ketamine + Placebo (Experimental): Subjects in this arm will receive (1) intravenous ketamine treatment once a week for 4 weeks (a total of 4 infusions) with a follow-up of 4 weeks and (2) intramuscular placebo once a month (a total of 2 injections).
  Interventions: Drug: Ketamine + Placebo
- Placebo (psychoactive placebo midazolam) + Placebo (Placebo Comparator): Subjects in this arm will receive (1) intravenous placebo treatment (psychoactive placebo midazolam) once a week for 4 weeks (a total of 4 infusions) with a follow-up of 4 weeks and (2) intramuscular placebo once a month (a total of 2 injections).
  Interventions: Drug: Placebo (psychoactive placebo midazolam) + Placebo

INTERVENTIONS:
Drug: Ketamine + Naltrexone — Subjects in this arm will receive (1) intravenous ketamine (0.5 mg/kg) once a week for 4 weeks (a total of 4 infusions) and (2) intramuscular naltrexone (380 mg) once a month (a total of 2 injections).
  Arms: Ketamine + Naltrexone
Drug: Ketamine + Placebo — Subjects in this arm will receive (1) intravenous ketamine (0.5 mg/kg) once a week for 4 weeks (a total of 4 infusions) and (2) intramuscular placebo once a month (a total of 2 injections).
  Arms: Ketamine + Placebo
Drug: Placebo (psychoactive placebo midazolam) + Placebo — Subjects in this arm will receive (1) intravenous psychoactive placebo midazolam (0.045 mg/kg) once a week for 4 weeks (a total of 4 infusions) and (2) intramuscular placebo once a month (a total of 2 injections).
  Arms: Placebo (psychoactive placebo midazolam) + Placebo

SUMMARY:
The investigators will compare 3 treatment groups (ketamine plus naltrexone vs. ketamine alone vs. placebo) for treating major depressive disorder (MDD) and alcohol use disorder (AUD) in an 8-week randomized, double-blind, placebo-controlled, between-subjects trial. First, prior to the double-blind trial, the investigators will conduct an open-label trial that will include 5 patients with comorbid MDD and AUD to test safety and efficacy of repeated ketamine treatment (0.5 mg/kg; once a week for 4 weeks; a total of 4 ketamine infusions) with a follow-up of 4 weeks. Second, after reviewing the safety and efficacy of repeated ketamine treatment from the open-label trial, the investigators will conduct an 8-week, randomized, double-blind, placebo-controlled trial that will include 60 patients with comorbid MDD and AUD to test safety and efficacy of repeated ketamine treatment (0.5 mg/kg; once a week for 4 weeks; a total of 4 ketamine infusions) plus naltrexone with a follow-up of 4 weeks. The 4-month follow-up session will also occur.

ELIGIBILITY:
Inclusion Criteria:

* Male or female veterans and civilians, 21-65 years old
* Current major depressive disorder without psychotic features by DSM-5 (antidepressant regimens can be allowed and changed during the trial)
* Montgomery-Asberg Depression Rating Scale (MADRS) 20 or higher
* A minimum of 4 of 11 current alcohol use disorder symptoms by DSM-5
* Heavy drinking at least 4 times in the past month ('heavy drinking' defined as 5 standard drinks per day for men and 4 standard drinks per day for women
* Able to provide written informed consent

Exclusion Criteria:

* Current substance use disorder by DSM-5 in the past 3 months (except alcohol, tobacco, or cannabis)
* Current or past history of psychotic features or psychotic disorder
* Current dementia
* Current uncontrolled hypertension (systolic BP > 170 mm Hg or diastolic BP > 100 mm Hg)
* Unstable medical condition or allergy to ketamine, midazolam, naltrexone, or lorazepam---clinically determined by a physician
* Imminent suicidal or homicidal risk
* Pregnant or nursing women, positive pregnancy test, or inadequate birth control methods in women of childbearing potential
* Positive opioid or illicit drug screen test (except marijuana)
* Opioid use within 10 days prior to study medication (injectable naltrexone) or risks for opioid use during the study
* Liver enzymes that are three times higher than the upper limit of normal
* Current use of benzodiazepine
* Acute narrow-angle glaucoma
* Severe sleep apnea---clinically determined by a physician

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gihyun Yoon, MD, Principal Investigator — VA Connecticut Healthcare System West Haven Campus, West Haven, CT
Locations (1):
- VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Analytic Code

REFERENCES:
- [Derived] Yoon G, Pittman B, Ralevski E, Petrakis IL, Krystal JH. Antidepressant efficacy of ketamine plus naltrexone for major depression comorbid with alcohol use disorder: a randomized controlled trial. Int J Neuropsychopharmacol. 2025 Aug 1;28(8):pyaf056. doi: 10.1093/ijnp/pyaf056. PMID 40795937

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ketamine + Naltrexone | Ketamine + Placebo | Placebo (Psychoactive Placebo Midazolam) + Placebo
Started | 22 | 21 | 22
Completed | 16 | 10 | 15
Not Completed | 6 | 11 | 7

BASELINE CHARACTERISTICS:
Population: Subjects receiving at least one infusion were analyzed
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine + Naltrexone | Ketamine + Placebo | Placebo (Psychoactive Placebo Midazolam) + Placebo | Total
Number analyzed (Participants) | 20 | 19 | 19 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Subjects receiving at least one infusion were analyzed
  years | 44.1 (13.7) | 50.0 (10.1) | 41.9 (13.5) | 45.3 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Subjects receiving at least one infusion treatment were analyzed.
  Participants
    Female | 4 | 4 | 5 | 13
    Male | 16 | 15 | 14 | 45
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Subjects receiving at least one infusion treatment were analyzed.
  Participants
    Race/Ethnicity: White | 18 | 14 | 7 | 39
    Race/Ethnicity: Black | 0 | 3 | 5 | 8
    Race/Ethnicity: Hispanic or Latino | 2 | 1 | 5 | 8
    Race/Ethnicity: Other | 0 | 1 | 2 | 3
Montgomery-Åsberg Depression Rating Scale (MADRS) score, mean (SD) [Mean (Standard Deviation); unit: units on a scale] — Montgomery-Åsberg Depression Rating Scale (MADRS):
  The total range: 0 - 60. Higher MADRS scores indicate a worse outcome (i.e., severe depression). Population: Subjects receiving at least one infusion treatment were analyzed.
  units on a scale | 27.8 (6.0) | 30.3 (6.1) | 30.3 (7.1) | 29.4 (6.4)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 50% or Greater Improvement in MADRS Scores From Baseline
Description: Our primary analysis (severity of depression) was to compare the proportions of subjects with clinical response in symptoms of major depressive disorder (response defined as a 50% or greater improvement from baseline in Montgomery-Asberg Depression Rating Scale (MADRS) scores) at the end-of-treatment time point (Day 21, after 4th infusion, T+240 minutes).
Time Frame: Day 21 (after 4th infusion, 240 minutes)
Population: Subjects who completed the outcome measure on Day 21 (after 4th infusion, 240 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine + Naltrexone | Ketamine + Placebo | Placebo (Psychoactive Placebo Midazolam) + Placebo
Number analyzed (Participants) | 16 | 11 | 15
Participants | 15 | 9 | 13

2. Primary Outcome: Rate of Complete Abstinence From Alcohol
Description: Alcohol consumption was measured using the Time Line Follow Back (TLFB) method. The rates of complete abstinence from alcohol across visits 3 (day 0) through visit 7 (day 28) were compared among the three study groups.
Time Frame: Day 28
Population: The total number of participants analyzed is inconsistent with the total number of participants reported in the same arm in the Participant Flow---because there is a lot of missing data in the TLFB.
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine + Naltrexone | Ketamine + Placebo | Placebo (Psychoactive Placebo Midazolam) + Placebo
Number analyzed (Participants) | 11 | 12 | 13
Participants | 3 | 6 | 2

ADVERSE EVENTS:
Time Frame: During the study period (8 weeks)
Description: Adverse events were collected using the Systematic Assessment for Treatment Emergent Effects (SAFTEE) method.
Arm/Group | Ketamine + Naltrexone | Ketamine + Placebo | Placebo (Psychoactive Placebo Midazolam) + Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 14/20 | 11/19 | 14/19
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ketamine + Naltrexone (N=20) | Ketamine + Placebo (N=19) | Placebo (Psychoactive Placebo Midazolam) + Placebo (N=19)
Blurred or double vision (General disorders) | 2 | 0 | 0
Chest pain, tightness, or discomfort (General disorders) | 0 | 1 | 3
General confusion (General disorders) | 1 | 0 | 0
Confusion as to time, place, person (General disorders) | 1 | 0 | 1
Cough (General disorders) | 3 | 2 | 6
Difficult, troubled breath or shortness of breath (General disorders) | 1 | 1 | 1
Difficult, burning, pain, frequent urge to urinate (General disorders) | 1 | 1 | 2
Difficulty with swallowing (General disorders) | 1 | 1 | 0
General dizziness (General disorders) | 2 | 1 | 1
Dizziness, faintness, lightheadedness upon rising (General disorders) | 2 | 1 | 3
Dream-like state (General disorders) | 1 | 2 | 2
Fast, slow, irregular heartbeat (General disorders) | 1 | 1 | 0
Flushing or redness of skin (General disorders) | 2 | 1 | 2
Irregular, fast, slow, or shallow breathing (General disorders) | 0 | 1 | 1
Itching (General disorders) | 1 | 2 | 2
Loss of appetite (General disorders) | 3 | 1 | 3
Nausea (General disorders) | 3 | 2 | 3
Pain at IV site (General disorders) | 2 | 2 | 1
Pale or blue lips, fingernails, skin (General disorders) | 1 | 0 | 0
Puffiness or swelling of eyelids or eyes (General disorders) | 3 | 0 | 1
Puffiness or swelling around eyes, face, lips, tongue (General disorders) | 2 | 0 | 1
Seeing, hearing, feeling things that are not there (General disorders) | 1 | 0 | 1
Skin rash (General disorders) | 1 | 0 | 0
Sweating (General disorders) | 3 | 1 | 3
Unusually warm skin (General disorders) | 2 | 1 | 1
Unusual excitement, nervousness, restlessness (General disorders) | 1 | 3 | 3
Unusual tiredness or weakness (General disorders) | 0 | 3 | 7
Vomiting (General disorders) | 1 | 0 | 2
Weight loss (General disorders) | 4 | 1 | 1
Headache (General disorders) | 4 | 1 | 6
Drowsiness (General disorders) | 2 | 2 | 6
Anxiety (General disorders) | 4 | 4 | 6
Tiredness (General disorders) | 4 | 2 | 6
Breast Pain (General disorders) | 1 | 1 | 0
Painful menstrual periods (General disorders) | 1 | 2 | 0
Missed menstrual periods (General disorders) | 2 | 1 | 0
Excessive menstrual bleeding (General disorders) | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-29): https://cdn.clinicaltrials.gov/large-docs/27/NCT02461927/Prot_SAP_000.pdf